CLINICAL TRIAL: NCT04731805
Title: "Moving On" - A Randomized Controlled Trial for Acceptability and Feasibility of an Early Physical Therapy Education Intervention for Breast Cancer Surgical Candidates
Brief Title: Moving On - An RCT to Test Physical Therapy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Ann Marie Flores, Assistant Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-04-17
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, longitudinal and prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moving On After Breast Cancer - Intervention Arm (Experimental): Participants are randomized to the intervention arm after their breast cancer diagnosis (but before cancer surgery) and baseline measurements (T0) are taken. They are followed up again at 2 weeks after their breast cancer surgery (T1), and again at 3 months after surgery (T2). Participants are given the patient education materials (booklet, therapeutic exercise DVD, small ball, range of motion wand). The research assistant orients the participant to the education materials and summarizes each section of the booklet. The research assistant also teaches the participant how to do the therapeutic exercises in the booklet. All participants in the intervention also receive usual care.
  Interventions: Behavioral: Moving On After Breast Cancer
- Usual Care (No Intervention): Participants are randomized to the usual care arm after their breast cancer diagnosis (but before cancer surgery) and baseline measurements (T0) are taken. They are followed up again at 2 weeks after their breast cancer surgery (T1), and again at 3 months after surgery (T2). Usual care consists of pre-operative testing, pre-operative nursing education on care of the surgical incision and pain management followed by breast cancer surgery.

INTERVENTIONS:
Behavioral: Moving On After Breast Cancer — Patient education intervention that is evidence-based, physical therapy, patient & family centered through the use of face to face instruction, a booklet, and therapeutic exercise DVD. The education materials are designed to deliver information on short term, long term, and late physical and functional effects of breast cancer treatment and given to breast cancer survivors before beginning cancer treatment. The education materials are designed to be used before, during, and after breast cancer treatment.
  Other Names: Intervention arm
  Arms: Moving On After Breast Cancer - Intervention Arm

SUMMARY:
The purpose of this study is to test the acceptability, feasibility and explore the possible effects of an early physical therapy education intervention for breast cancer survivors.

DETAILED DESCRIPTION:
This study uses a randomized controlled and longitudinal study design. We will compare two groups - an intervention group and a control group - to test the effects of an early physical therapy education intervention for breast cancer survivors who are candidates for breast cancer surgery. Because of the nature of the intervention (patient early education with 1:1 discussion of educational materials) we will be unable to introduce blinding of the participant as well as the staff.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with unilateral breast cancer
* Candidate for breast cancer surgery as first line of cancer treatment
* Undergo breast cancer surgery at Brigham and Woman's Hospital, Boston, Massachusetts
* Female
* English speaking
* Greater than or equal to 21 years old

Exclusion Criteria:

* Previous history of breast cancer and/or recurrent/metastatic disease
* Receiving neoadjuvant chemotherapy treatment
* Bilateral breast cancer
* History of shoulder impairments or severe upper quarter scarring
* Pregnancy
* Central nervous system damage
* Dementia
* History of other previous cancers (except non-melanoma skin)
* Systemic medical conditions (e.g.: fibromyalgia, rheumatoid arthritis, etc.)
* Amputation of either upper extremity

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05-23 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2015-05-22 (Actual)

PRIMARY OUTCOMES:
Change in active shoulder range of motion | 3 months
  Active shoulder range of motion is measured with a standard goniometer in degrees. Change from baseline to 3 months for shoulder flexion, extension, abduction, and internal and external ranges are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Flores, PhD, Principal Investigator — Northeastern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warren C. Physical therapy intervention suggestions for women following breast cancer surgery. Journal of Women's Health Physical Therapy. 2005;29(1):21-24.
- [Background] Mustian KM, Peppone L, Darling TV, Palesh O, Heckler CE, Morrow GR. A 4-week home-based aerobic and resistance exercise program during radiation therapy: a pilot randomized clinical trial. J Support Oncol. 2009 Sep-Oct;7(5):158-67. PMID 19831159
- [Background] McNeely ML, Campbell K, Ospina M, Rowe BH, Dabbs K, Klassen TP, Mackey J, Courneya K. Exercise interventions for upper-limb dysfunction due to breast cancer treatment. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD005211. doi: 10.1002/14651858.CD005211.pub2. PMID 20556760
- [Background] Torres Lacomba M, Yuste Sanchez MJ, Zapico Goni A, Prieto Merino D, Mayoral del Moral O, Cerezo Tellez E, Minayo Mogollon E. Effectiveness of early physiotherapy to prevent lymphoedema after surgery for breast cancer: randomised, single blinded, clinical trial. BMJ. 2010 Jan 12;340:b5396. doi: 10.1136/bmj.b5396. PMID 20068255
- [Background] Schmitz KH, Ahmed RL, Troxel A, Cheville A, Smith R, Lewis-Grant L, Bryan CJ, Williams-Smith CT, Greene QP. Weight lifting in women with breast-cancer-related lymphedema. N Engl J Med. 2009 Aug 13;361(7):664-73. doi: 10.1056/NEJMoa0810118. PMID 19675330